CLINICAL TRIAL: NCT00639210
Title: BREAST CANCER AND EXERCISE BREX: A Multicenter Phase III Open Randomised Trial of the Efficacy of Exercise in the Prevention of Long-term Adverse Effects of Adjuvant Treatments and Breast Cancer Recurrences in Women With Primary Breast Cancer.
Brief Title: BREAST CANCER AND EXERCISE
Acronym: BREX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Finnish Breast Cancer Group (Other)
Responsible Party: Riikka Huovinen, Finnish Brest Cancer Group
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Protocol number FBCSG-01-2004
Record Dates: First submitted 2008-03-14; First posted 2008-03-20 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Prevent Osteoporosis and Osteoporotic Fractures; Improve Quality of Life; Improve Weight Control, and Muscular and Cardiovascular Fitness; Help the Patients to Return to Working Life; Reduce the Risk of Breast Cancer Recurrence; Reduce All-cause Mortality in Patients With Primary Breast Cancer
Keywords: breast cancer; exercise; osteoporosis; fracture; quality of life
MeSH Terms: conditions — Osteoporotic Fractures; Breast Neoplasms; Motor Activity; Osteoporosis; Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Other): Supervised training is organised for the exercise group once a week in groups of 10 to 15 subjects. The training is guided by an experienced physical therapist.
  Interventions: Other: supervised training
- B (No Intervention)

INTERVENTIONS:
Other: supervised training — Design: supervised training is organised for the exercise group once a week in groups of 10 to 15 subjects. The training is guided by an experienced physical therapist.Content: The supervised training of the exercise group consists of two different classes alternating at four week periods; step aerobics class and circuit training class. The 60-minute aerobics and circuit training classes also include warming-up and cooling-down periods both lasting 10-15 minutes.
  Arms: A

SUMMARY:
A Finnish Breast Cancer Group Study (BREX 01-2004). A multicenter phase III open randomised trial of the efficacy of exercise in the prevention of long-term adverse effects of adjuvant treatments and breast cancer recurrences in women with primary breast cancer. The aim of the study is to investigate whether regular exercise training could reduce the long-term side effects of adjuvant treatments of primary breast cancer and improve quality of life and well being.

DETAILED DESCRIPTION:
A multicenter phase III open randomised trial of the efficacy of exercise in the prevention of long-term adverse effects of adjuvant treatments and breast cancer recurrences in women with primary breast cancer. The aim of the study is to investigate whether regular exercise training could reduce the long-term side effects of adjuvant treatments of primary breast cancer and improve quality of life and well being. Large controlled prospective studies are needed to confirm the preliminary findings of exercises benefits in cancer patients, and to investigate the type, the frequency, intensity and tolerability of exercise training in cancer patients, before any clinical recommendations can be given. Prevention of osteoporosis, improvement of weight control, and muscular and cardiovascular fitness is been waited. The second aim of the study is to investigate, whether regular exercise training reduces the risk of breast cancer recurrence, prevents other diseases and reduce all-cause mortality and is cost effective in women with primary breast cancer.

ELIGIBILITY:
Inclusion Criteria: Histologically proven invasive breast cancer T1-4N0-3M0, pre- or postmenopausal breast cancer patient treated with adjuvant chemotherapy or radiotherapy within 4 months or patient who has started adjuvant endocrine therapy (antiestrogens, aromatase inhibitors, LHRH agonists, or combinations) no later than 4 months earlier,age from 35 to 68 years,signed informed consent prior to beginning protocol specific procedures

Exclusion Criteria:

* Prior malignancy except basal cell carcinoma or in situ cervix carcinoma
* Male gender
* Haematogenous metastases (M1)
* No systemic adjuvant therapy
* Postmenopausal women treated with antiestrogens, tamoxifen or toremifene, adjuvant treatment only (+/- radiotherapy)
* Pregnancy or recent lactation (< 1 year)
* Severe cardiac disease (New York Heart Association class III or greater), myocardial infarction within 12 months, uncontrolled hypertension
* Verified osteoporosis (proximal femur or lumbar spine t-score < -2.5 or fracture without trauma)
* Concomitant medications affecting calcium and bone metabolism such as bisphosphonates, calcitonin, PTH, SERMs, oral corticosteroids (over 6 months), anticonvulsants (fenytoin, carbamazepine) and prolonged heparin therapy
* Other diseases affecting calcium and bone metabolism such as hyperthyroidism, newly diagnosed hypothyroidism, primary hyperparathyroidism, renal failure, chronic hepatic diseases, organ transplant, Cushing's syndrome, rheumatoid arthritis, chronic bowel diseases such as celiac disease, Chron disease or history of total ventricular resection
* Other serious illness or medical condition, which could be contraindication for exercise
* Patients not capable of training (severe knee arthrosis, severe ligamental or cartilage injuries at lower extremities)
* Residence more than one hour from the exercise centre
* Competitive athlete

Ages: 35 Years to 68 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 573 (Actual)
Dates: Start 2005-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The aim of the study is to investigate whether regular exercise after adjuvant treatments of breast cancer could prevent osteoporosis and improve quality of life. | 1-10 years

SECONDARY OUTCOMES:
Fitness and weight control, number of falls and fractures, breast cancer recurrence. | 1-10 years

CONTACTS AND LOCATIONS:
Overall Officials: Tiina Saarto, MD, PhD, Principal Investigator — Helsinki University Central Hospital, Department of Oncology
Locations (1):
- Helsinki University Central Hospital, Department of Oncology, Helsinki, Finland

REFERENCES:
- [Derived] Blomqvist C, Vehmanen L, Kellokumpu-Lehtinen PL, Huovinen R, Ruohola J, Penttinen H, Sievanen H, Nikander R, Utriainen M, Saarto T. Long-term effects of aromatase inhibitor withdrawal on bone mineral density in early breast cancer patients: 10-year follow-up results of the BREX study. Breast Cancer Res Treat. 2024 Jul;206(1):57-65. doi: 10.1007/s10549-024-07252-7. Epub 2024 Apr 1. PMID 38561578
- [Derived] Poikonen-Saksela P, Kolokotroni E, Vehmanen L, Mattson J, Stamatakos G, Huovinen R, Kellokumpu-Lehtinen PL, Blomqvist C, Saarto T. A graphical LASSO analysis of global quality of life, sub scales of the EORTC QLQ-C30 instrument and depression in early breast cancer. Sci Rep. 2022 Feb 8;12(1):2112. doi: 10.1038/s41598-022-06138-2. PMID 35136160
- [Derived] Penttinen HM, Saarto T, Kellokumpu-Lehtinen P, Blomqvist C, Huovinen R, Kautiainen H, Jarvenpaa S, Nikander R, Idman I, Luoto R, Sievanen H, Utriainen M, Vehmanen L, Jaaskelainen AS, Elme A, Ruohola J, Luoma M, Hakamies-Blomqvist L. Quality of life and physical performance and activity of breast cancer patients after adjuvant treatments. Psychooncology. 2011 Nov;20(11):1211-20. doi: 10.1002/pon.1837. Epub 2010 Sep 27. PMID 20878646